CLINICAL TRIAL: NCT03882723
Title: Carbon Dioxide (CO2) Clearance From Various Face Masks in Normal Volunteers at Various Level of Expiratory Positive Airway Pressure (EPAP) When Using a Non-Invasive Positive Pressure Ventilation (NIPPV)
Brief Title: Noninvasive Ventilation Masks Carbon Dioxide Clearance in Normal Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORA: 18011502-IRB01
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: CO2 Clearance; Mask Comfort; Rebreathing Exhaled Gas
MeSH Terms: interventions — Noninvasive Ventilation; Ventilators, Mechanical

STUDY DESIGN:
Intervention Model Description: randomized crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Randomized Crossover Trial with 4 NIV Masks (Experimental): Order of the masks (BiTrac MaxShield™ with standard elbow, BiTrac™ Full Face with standard elbow, Respironics PerforMax with standard elbow, and Respironics AF531 with standard elbow) were randomly chosen. Investigators randomly assigned all masks for paper raffling from container. All subjects performed 20 minutes on each mask followed by 5 minutes wash out between masks. EPAP levels will be 0, 2, 4, & 5 (5 minutes for each level) while IPAP remains at 5 higher than EPAP. FiCO2 and EtCO2 were collected at 4:00, 4:30 and 5:00 minute mark for each EPAP level. Also, subjective mask comfort was assessed via visual analog scale (VAS) with 1 referring to least comfortable and 5 being the most comfortable after 5 each EPAP setting.
  Interventions: Device: Evaluated 4 masks used for NIV with mechanical ventilators

INTERVENTIONS:
Device: Evaluated 4 masks used for NIV with mechanical ventilators — Order of the masks (BiTrac MaxShield™ with standard elbow, BiTrac™ Full Face with standard elbow, Respironics PerforMax with standard elbow, and Respironics AF531 with standard elbow) were randomly chosen. Investigators randomly assigned all masks for paper raffling from container. All subjects performed 20 minutes on each mask followed by 5 minutes wash out interval between masks. EPAP levels will be 0, 2, 4, & 5 (5 minutes for each level) while IPAP remains at 5 higher than EPAP. FiCO2 and EtCO2 were collected at 4:00, 4:30 and 5:00 minute mark for each EPAP level. Also, subjective mask comfort was assessed via visual analog scale (VAS) with 1 referring to least comfortable and 5 being the most comfortable after 5 each EPAP setting.

SUMMARY:
This study will be a randomized crossover trial that will be conducted at Rush University. The study will be conducted with 20 healthy volunteers who will be placed on ICU ventilator operating in the NIPPV mode. All subjects will perform 15 minutes of breathing on NIPPV on each mask of the 4 different masks (2 oronasal and 2 full face masks) that are randomly selected. Breathing through each mask will be followed by a 5- minute wash out period between masks. End tidal Carbon Dioxide (EtCO2) will be sampled nasal/oral. Different levels of EPAP will be set and CO2 clearance will be monitored. Additionally, subjective mask comfort will be assessed via visual analog scale (VAS) with 1 referring to least comfortable and 5 being the most comfortable.

DETAILED DESCRIPTION:
This study will be a randomized crossover trial that will be conducted at Rush University. Normal volunteers will be recruited from Rush University Medical Centers. Volunteers will be screened with inclusion and exclusion criteria and an informed consent is required in order for them to participate.

Also, initial baseline vital signs (heart rate, blood pressure, respiratory rate, and oxygen saturation) will be obtained. EtCO2 will be obtained at baseline and periodically using an oral/nasal sample line with the CapnostreamTM 20p monitor (Medtronic, Minneapolis, MN). The study will use a double limb circuit ICU ventilator Puritan Bennett™ (Medtronic, Dublin, Ireland).

Investigators will evaluate 4 NIPPV masks (2 oronasal masks and 2 full face masks). Oronasal masks will be labeled as group A and numbered as A1 and A2; while full face masks will be labeled group B and numbered as B1 and B2. Order of the masks will be randomly chosen in two steps. First steps will be choosing A or B then randomly assign mask in each of these groups. Investigators will randomly assign mask in group A or B by drawing an initial mask from the group and then continue the sequence of masks from that point. For example, investigators randomly chose group A, then randomly chose A2, the sequence will be A2, A1. Then Investigators would randomly choose B2, then the sequence would be B2, B1. All subjects will perform 15 minutes on each mask followed by 5 minutes wash out interval between masks. EPAP levels will be 0, 2, 4, & 5 while IPAP remains at 5 higher than EPAP. EtCO2 will be collected at 4:00, 4:30 and 5:00 minute mark. These three measures should differ by less than 20% of their average. Also, subjective mask ORA: 18011502-IRB01 Date IRB Approved: 3/30/2018 Amendment Date: 5/11/2018 comfort will be assessed via visual analog scale (VAS) with 1 referring to least comfortable and 5 being the most comfortable after 5 each EPAP setting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects greater than 18 years old.

Exclusion Criteria:

* Prior history of NIPPV as a patient.
* Facial surgery or deformity
* Ear infection
* History of pulmonary or cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Vines, PhD, Study Chair — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomized crossover trial so each participate used all four masks (BiTrac MaxShield™ with standard elbow, BiTrac™ Full Face with standard elbow, Respironics PerforMax with standard elbow, and Respironics AF531 with standard elbow).
Groups:
- Randomized Crossover Trial With 4 NIV Masks: Order of the 4 masks (BiTrac MaxShield™ with standard elbow, BiTrac™ Full Face with standard elbow, Respironics PerforMax with standard elbow, and Respironics PerforMax with standard elbow) were randomly chosen. Investigators randomly assigned all masks for paper raffling from container. All subjects performed 20 minutes on each mask followed by 5 minutes wash out interval between masks. EPAP levels will be 0, 2, 4, & 5 (5 minutes for each level) while IPAP remains at 5 higher than EPAP. FiCO2 and EtCO2 were collected at 4:00, 4:30 and 5:00 minute mark for each EPAP level. Also, subjective mask comfort was assessed via visual analog scale (VAS) with 1 referring to least comfortable and 5 being the most comfortable after 5 each EPAP setting.
  Evaluated masks used for NIV with mechanical ventilators: Order of the masks were randomly chosen. Investigators randomly assigned all masks for paper raffling from container. All subjects performed 20 minutes on each mask followed by 5 minutes wash out interval between masks. EPAP levels will be 0, 2, 4, & 5 (5 minutes for each level) while IPAP remains at 5 higher than EPAP. FiCO2 and EtCO2 were collected at 4:00, 4:30 and 5:00 minute mark for each EPAP level. Also, subjective mask comfort was assessed via visual analog scale (VAS) with 1 referring to least comfortable and 5 being the most comfortable after 5 each EPAP setting.
Period: Overall Study
Arm/Group | Randomized Crossover Trial With 4 NIV Masks
Started | 8
BiTrac Max Shield | 8
BiTrac™ Full Face | 8
Respironics PerforMax | 8
Respironics AF531 | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Crossover Trial With 4 NIV Masks: Order of the masks (BiTrac MaxShield™ with standard elbow, BiTrac™ Full Face with standard elbow, Respironics PerforMax with standard elbow, and Respironics PerforMax with standard elbow) were randomly chosen. Investigators randomly assigned all masks for paper raffling from container. All subjects performed 20 minutes on each mask followed by 5 minutes wash out interval between masks. EPAP levels will be 0, 2, 4, & 5 (5 minutes for each level) while IPAP remains at 5 higher than EPAP. FiCO2 and EtCO2 were collected at 4:00, 4:30 and 5:00 minute mark for each EPAP level. Also, subjective mask comfort was assessed via visual analog scale (VAS) with 1 referring to least comfortable and 5 being the most comfortable after 5 each EPAP setting.
  Evaluated masks used for NIV with mechanical ventilators: Order of the masks were randomly chosen. Investigators randomly assigned all masks for paper raffling from container. All subjects performed 20 minutes on each mask followed by 5 minutes wash out interval between masks. EPAP levels will be 0, 2, 4, & 5 (5 minutes for each level) while IPAP remains at 5 higher than EPAP. FiCO2 and EtCO2 were collected at 4:00, 4:30 and 5:00 minute mark for each EPAP level. Also, subjective mask comfort was assessed via visual analog scale (VAS) with 1 referring to least comfortable and 5 being the most comfortable after 5 each EPAP setting.
Arm/Group | Randomized Crossover Trial With 4 NIV Masks
Number analyzed (Participants) | 8
Age, Customized [Count of Participants; unit: Participants] — Greater than 18 years of age
  Participants
    greater than 18 | 8
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: This data was not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
No history of pulmonary or cardiac disease [Count of Participants; unit: Participants] — Participants asked if they had a history of pulmonary or cardiac disease.
  Participants | 8
No current ear infection [Count of Participants; unit: Participants] — Participants were asked if they had an ear infection.
  Participants | 8
No history of use of noninvasive ventilation [Count of Participants; unit: Participants] — Participants were asked if they had used noninvasive ventilation before.
  Participants | 8
no facial surgery or deformity that would interfere with the mask seal. [Count of Participants; unit: Participants] — participants were observed for face deformities or surgery that would interfere with the mask seal.
  Participants | 8

OUTCOME MEASURES:

1. Primary Outcome: Carbon Dioxide Clearance From the Masks
Description: Measured the percentage of CO2 being re-breathed or inspired using a nasal cannula and sidestream end-tidal CO2 monitor.
Time Frame: 5 min
Population: The study protocol and statistical analysis planned to have this outcome measure be analyzed and reported per PEEP level, not per intervention. There were 8 participants and 4 masks, making 32 unique measures for each PEEP level. This pilot project aimed to identify that CO2 rebreathing existed when using a dual limb circuit. Individual mask data may misrepresent the issue and be inappropriately used for marketing purposes.
Measure: Median (Inter-Quartile Range); unit: percentage of CO2 inspired
Groups:
- PEEP 0: A PEEP of 0 cmH2O was applied to the masks.
- PEEP 2: A PEEP of 2 cmH2O was applied to the masks.
- PEEP 4: A PEEP of 4 cmH2O was applied to the masks.
- PEEP 5: A PEEP of 5 cmH2O was applied to the masks.
Arm/Group | PEEP 0 | PEEP 2 | PEEP 4 | PEEP 5
Number analyzed (Participants) | 8 | 8 | 8 | 8
percentage of CO2 inspired | 1.83 [0.66 to 4] | 1 [0.33 to 2.66] | 0.49 [0 to 1.92] | 0 [0 to 0.92]

2. Secondary Outcome: Leak (L/Min)
Description: Amount of leak measured by the ventilator.
Time Frame: 5 min
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Liters per minute
Groups:
- PEEP 0; PEEP 4: All masks at a PEEP of 0 cmH2O
- PEEP 2: All masks at a PEEP of 2 cmH2O
- PEEP 5: All masks at a PEEP of 5 cmH2O
Arm/Group | PEEP 0 | PEEP 2 | PEEP 4 | PEEP 5
Number analyzed (Participants) | 8 | 8 | 8 | 8
Liters per minute | 22 [15 to 30] | 30 [25 to 40] | 36 [27 to 41] | 41 [33 to 47]

3. Secondary Outcome: Tidal Volume
Description: Tidal volume measured by the ventilator.
Time Frame: 5 minutes
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: milliliters
Arm/Group | PEEP 0 | PEEP 2 | PEEP 4 | PEEP 5
Number analyzed (Participants) | 8 | 8 | 8 | 8
milliliters | 636 [503 to 892] | 646 [496 to 908] | 637 [498 to 938] | 701 [481 to 968]

4. Secondary Outcome: Respiratory Rate (BPM)
Description: The ventilator measured the subjects' respiratory rates.
Time Frame: 5 minutes
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: breaths per minute
Arm/Group | PEEP 0 | PEEP 2 | PEEP 4 | PEEP 5
Number analyzed (Participants) | 8 | 8 | 8 | 8
breaths per minute | 13 [12 to 17] | 15 [12 to 17] | 15 [12 to 18] | 15 [13 to 18]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during data collection which was approximately 1.5 hours.
Description: The study would be stopped if subjects' HR changed by 20% from baseline for more than 1 min and/or complained of shortness of breath.
Groups:
- Randomized Crossover Trial With 4 NIV Masks: Order of the 4 masks were randomly chosen. Investigators randomly assigned all masks for paper raffling from a container. All subjects performed 20 minutes on each mask followed by 5 minutes wash out between masks. EPAP levels will be 0, 2, 4, & 5 (5 minutes for each level), while IPAP remains at 5 higher than EPAP. FiCO2 and EtCO2 were collected at 4:00, 4:30 and 5:00 minute mark for each EPAP level.
  The study protocol and statistical analysis planned to have all outcome measures and adverse events be analyzed and reported per PEEP level, not per intervention.
Arm/Group | Randomized Crossover Trial With 4 NIV Masks
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT03882723/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT03882723/ICF_001.pdf